CLINICAL TRIAL: NCT06285084
Title: Deep Learning ECG Evaluation and Clinical Assessment for Competitive Sport Eligibility
Acronym: VALETUDO
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: VALETUDO Trial (L4195)
Record Dates: First submitted 2024-02-05; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Sports Cardiology; Preventive Cardiology; Electrocardiogram; Artificial Intelligence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training Cohort: 455 Athletes already evaluated for sports participation clearance, whom ECG and clinical evaluation (cleared - not cleared for competitive sports participation) will be fed into the DL model
- Validation Cohort: 76 Athletes evaluated using standard sports eligibility clearance tests and our DL model

SUMMARY:
The goal of this observationl study is to evaluate the possibility of building a Deep Learning (DL) model capable of analyzing electrocardiographic traces of athletes and providing information in the form of a probability stratification of cardiovascular disease.

Researchers will enroll a training cohort of 455 participants, evaluated following standard clinical practice for eligibility in competitive sports. The response of the clinical evaluation and ECG traces will be recorded to build a DL model.

Researchers will subsequently enroll a validation cohort of 76 participants. ECG traces will be analyzed to evaluate the accuracy of the model to discriminate participants cleared for sports eligibility versus participants who need further medical tests

DETAILED DESCRIPTION:
The goal of this observationl study is to evaluate the possibility of building a Deep Learning (DL) model capable of analyzing electrocardiographic traces of athletes and providing information in the form of a probability stratification of cardiovascular disease.

The DL model requires training to be calibrated. The project plans to conduct accuracy evaluations on the validation population (76 athletes) and training trials on a different dataset (455 athletes).

There will be an initial phase of system training. Athletes will be assessed according to current guidelines and the italian cardiological guidelines for competitive sports participation - COCIS, with the required diagnostic tests on a case-by-case basis. At the end of the cardiac evaluation, athletes can be classified as "fit" or "unfit" for competitive activity.

Participants will submit the ECGs of "fit" and "unfit" athletes, categorized into these two groups, to a deep learning algorithm to train the artificial intelligence system.

A population of consecutive athletes will then be recruited to form the validation set for the test. These athletes have indications for evaluation for the granting of competitive fitness, as indicated by the referring sports physicians. In this case as well, athletes in the validation set will be assessed according to guidelines and COCIS with appropriate tests on a case-by-case basis to evaluate fitness for competition.

Participants will subject the ECGs of the validation set athletes to the artificial intelligence model to assess accuracy, sensitivity, specificity, positive predictive value, negative predictive value, and AUC in discriminating athletes judged "fit" from those judged "unfit" for competitive activity after cardiac investigations.

ELIGIBILITY:
Inclusion Criteria:

* Athletes in need of cardiac or sports medical evaluation for the issuance of competitive eligibility.
* Enlisted athletes involved in sports like soccer or those with mixed or aerobic cardiovascular demands according to the COCIS 2017 classification.
* Aged 18 years or older but not exceeding 60 years.
* No history of cardiovascular disease.
* Signed Informed Consent.

Exclusion Criteria:

* Athletes engaging in skill-based sports as per the COCIS 2017 classification.
* High clinical probability of cardiovascular disease, such as typical angina or heart failure.
* Pregnancy and/or breastfeeding (confirmed through self-declaration).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adults requiring medical evaluation for competitive sports eligibility
Sampling Method: Non-Probability Sample
Enrollment: 531 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
DL model accuracy | From first medical evaluation with ECG until the final medical decision on competitive sports eligibility, up to 12 months
  The accuracy of the DL model in recognizing the ECGs of athletes deemed fit or unfit will be evaluated by comparing the results with those obtained from the assessment performed by the sports physician (gold standard).
  Participants will categorize the athletes into true positives, false positives, true negatives, and false negatives.
  To define the ability of the DL model to discriminate between ECGs of athletes deemed fit or unfit, the receiver operating characteristic (ROC) curve and the corresponding area under the curve (AUC) will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Galeazzi-Sant'Ambrogio, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: Undecided